CLINICAL TRIAL: NCT02687932
Title: Multicenter, Randomized, Double-blind, Active-controlled Study to Assess the Efficacy of LCZ696 Compared to Valsartan on Reduction of Mitral Regurgitation in Patients With Left Ventricular Dysfunction and Secondary Functional Mitral Regurgitation of Stage B and C
Brief Title: Pharmacological Reduction of Functional, Ischemic Mitral REgurgitation
Acronym: PRIME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Duk-Hyun Kang, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-0938
Record Dates: First submitted 2016-02-17; First posted 2016-02-22 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Mitral Valve Insufficiency; Left Ventricular Dysfunction
Keywords: Functional Mitral Regurgitation; Ischemic Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency; Ventricular Dysfunction, Left | interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LCZ696 (Experimental): LCZ696 for 12 months
  Interventions: Drug: LCZ696
- Valsartan (Active Comparator): Valsartan for 12 months
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: LCZ696
  Arms: LCZ696
Drug: Valsartan
  Arms: Valsartan

SUMMARY:
Functional MR is caused by adverse left ventricular remodeling after myocardial injury and associated with an increased incidence of heart failure and death. Because secondary functional MR usually develops as a result of LV dysfunction, diuretics, beta blockers, angiotensin-converting-enzyme (ACE) inhibitors or angiotensin receptor blockers (ARB), and aldosterone antagonists are given to patients with functional MR in line with the guidelines in the management of heart failure. However, functional MR appears to remain common despite use of these drugs and current medical treatment is usually insufficient for reducing MR or reversing the adverse LV remodeling. As LCZ696 is a dual-acting inhibitor of the renin-angiotensin-aldosterone system (RAAS) and neutral endopeptidase (NEP), LCZ696 has greater hemodynamic and neurohormonal effects than ARB alone. Investigators try to examine the hypothesis that LCZ696 is superior to ARB alone in improving functional MR in patients with LV dysfunction and functional MR.

DETAILED DESCRIPTION:
Functional ischemic mitral regurgitation (MR) has been reported to occur in up to 40% of patients after myocardial infarction, and the prevalence of functional MR is likely to increase with an aging population and improved survival rates for myocardial infarction. The presence of functional MR is associated with an increased incidence of heart failure and death, and patients with significant functional MR incur about a two-fold increase in the risk of mortality and about a four-fold increase in the risk of heart failure. Functional MR is caused by adverse left ventricular remodeling after myocardial injury with enlargement of the left ventricle (LV), apical and lateral displacement of papillary muscles, leaflet tethering and reduced closing forces. The leaflets are normal in secondary functional MR and the treatment is considerably different between functional and primary MR. Surgery is the only definitive therapy for primary severe MR and primary MR can usually be cured by surgical valve repair. However, surgical indications are unclear in severe functional MR, because outcomes after surgery for functional MR remain suboptimum. Operative mortality, long-term mortality and heart failure rates are still high in patients with severe functional MR despite surgical improvements. According to the current guidelines, mitral valve surgery may be considered only for severely symptomatic patients with severe secondary functional MR who have persistent symptoms despite optimal medical therapy for heart failure.

Because secondary functional MR usually develops as a result of LV dysfunction, diuretics, beta blockers, angiotensin-converting-enzyme (ACE) inhibitors or angiotensin receptor blockers (ARB), and aldosterone antagonists are given to patients with functional MR in line with the guidelines in the management of heart failure. However, functional MR appears to remain common despite use of these drugs and current medical treatment is usually insufficient for reducing MR or reversing the adverse LV remodeling. Persistence of functional MR due to the insufficient effectiveness of current medical treatment significantly increases morbidity and mortality, and compared with surgical or percutaneous revascularization, significantly higher mortality was observed in patients managed with medical therapy.

Quantitative assessment of MR is strongly recommended in the guidelines and the regurgitant volume and the effective regurgitant orifice area (EROA) of MR can be measured accurately and reproducibly by Doppler echocardiography. The EROA of MR has an important prognostic value in primary and secondary functional MR. Because functional MR carries an adverse prognosis with a graded relationship between MR severity and reduced survival, therapies that induce beneficial reverse remodeling of the LV and reduce MR, may improve survival. ACE inhibitors and ARBs could partially attenuate LV dilatation and remodeling after myocardial injury, but there are no published data from prospective trials regarding whether attenuation of remodeling by ACE inhibitors or ARBs reduces functional MR.

LCZ696 is a dual-acting inhibitor of the renin-angiotensin-aldosterone system (RAAS) and neutral endopeptidase (NEP). As LCZ696 offers the therapeutic advantages of concomitantly blocking both RAAS and NEP, LCZ696 was more effective in reducing the risk of death from cardiovascular causes or hospitalization for heart failure in patients with chronic heart failure than ACE inhibitor. Because NEP is involved in the metabolism of a number of vasoactive peptides such as natriuretic peptides, NEP inhibitor has vasodilating effects, facilitates sodium excretion and has profound effects on LV remodeling. Trials of hypertension and heart failure with a preserved ejection fraction also showed that LCZ696 had greater hemodynamic and neurohormonal effects than ARB alone. To date, there has been no proven pharmacological therapy to improve functional MR, and the development of medical therapy should be at the forefront of research considering the limited role of surgery in managing functional MR. Investigators hypothesize that LCZ696 is superior to ARB alone in improving functional MR in patients with LV dysfunction and functional MR via synergistic effects of NEP and RAAS inhibition on LV remodeling, and try to examine this hypothesis in a multicenter, double-blind, randomized comparison study using echocardiography.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must agree to the study protocol and provide written informed consent
2. Outpatients ≥ 20 years of age, male or female
3. Patients with secondary functional MR (stage B and C) and LV dysfunction

   * Symptoms due to coronary ischemia or heart failure may be present but symptoms due to MR should be absent
   * Normal mitral valve leaflets and chords
   * Regional or global wall motion abnormalities with mild or severe tethering of leaflet
   * ERO > 0.10 cm2
   * 25% < LV ejection fraction < 50%
4. Dyspnea of NYHA functional class II or III
5. Patients must be on stable, optimized dose of an ACE inhibitors or ARBs for at least 4 weeks prior to study entry

Exclusion Criteria:

1. History of hypersensitivity or allergy to the study drug, drugs of similar chemical classes, ARBs, or NEP inhibitors as well as known or suspected contraindications to the study drug
2. Known history of angioedema
3. Any evidence of structural mitral valve disease, including prolapse of mitral leaflets and rupture of chords or papillary muscles
4. Current acute decompensated heart failure or dyspnea of NYHA functional class IV
5. Medical history of hospitalization within 6 weeks
6. Symptomatic hypotension and/or a SBP < 100 mmHg at screening
7. Estimated GFR < 30 mL/min/1.73m2
8. Serum potassium > 5 mmol/L at screening
9. Evidence of hepatic disease as determined by any one of the following: AST or ALT values exceeding 2 x upper limit of normal (ULN) at screening visit (Visit 0), history of hepatic encephalopathy, history of esophageal varices, or history of portacaval shunt
10. Acute coronary syndrome, stroke, major CV surgery, PCI within 3 months
11. Planned coronary revascularization or mitral valve intervention within 1 year
12. Heart transplantation or implantation of cardiac resynchronization therapy
13. History of severe pulmonary disease
14. Significant aortic valve disease
15. Primary aldosteronism
16. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using a barrier method plus a hormonal method
17. Pregnant or nursing (lactating) women
18. Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the investigator, would preclude safe completion of the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-01-02 (Actual)

PRIMARY OUTCOMES:
Change of effective regurgitant orifice area (EROA) of functional mitral regurgitation from baseline to 12 months follow-up | 12 months

SECONDARY OUTCOMES:
Change of regurgitant volume from baseline to 12 months follow-up | 12 months
Change of left ventricular end-systolic volume from baseline to 12 months follow-up | 12 months
Change of left ventricular end-diastolic volume from baseline to 12 months follow-up | 12 months
Change of incomplete mitral leaflet closure area from baseline to 12 months follow-up | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Duk-Hyun Kang, M.D., Principal Investigator — Asan Medical Center
Locations (4):
- South Korea (4):
  - Inha University Hospital, Incheon
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Yonsei University Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kang DH, Park SJ, Shin SH, Hong GR, Lee S, Kim MS, Yun SC, Song JM, Park SW, Kim JJ. Angiotensin Receptor Neprilysin Inhibitor for Functional Mitral Regurgitation. Circulation. 2019 Mar 12;139(11):1354-1365. doi: 10.1161/CIRCULATIONAHA.118.037077. PMID 30586756